CLINICAL TRIAL: NCT00316563
Title: A Double-blind, Randomized, Placebo Controlled Clinical Trial to Evaluate the Efficacy of Orexigenic Therapy With Delta-9-tetrahydrocannabinol in Advanced Cancer Patients With Chemosensory Abnormalities - a Pilot Study
Brief Title: Orexigenic Therapy With Delta-9-tetrahydrocannabinol in Advanced Cancer Patients With Chemosensory Abnormalities - a Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alberta Health services (Other)
Collaborators: University of Alberta (Other)
Organization: AHS Cancer Control Alberta (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PS-8-0008
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2007-11

CONDITIONS: Cancer; Anorexia; Taste Disorders; Olfactory Disorders
Keywords: cannabinoids; taste disorders; olfaction disorders; cancer; palliative medicine; caloric intake; appetite; reward; tetrahydrocannabinol/therapeutic use; anorexia/drug therapy; quality of life; chemosensory changes/drug therapy
MeSH Terms: conditions — Neoplasms; Anorexia; Taste Disorders; Olfaction Disorders | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Marinol (Dronabinol)
- 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Marinol (Dronabinol) — Intervention description: Marinol (drug) is being used as an appetite stimulant for treatment of cancer-induced anorexia.
  Arms: 1
Other: Placebo
  Arms: 2

SUMMARY:
To investigate delta-9-tetrahydrocannabinol's (THC) ability to increase food intake and improve food enjoyment for advanced cancer patients with taste and/or smell (chemosensory) abnormalities.

DETAILED DESCRIPTION:
Appetite stimulants are the common treatment for cancer-induced anorexia. However, only 30% of advanced cancer patients respond and benefit from appetite stimulants, which may be due in part to sensory abnormalities, as a person who is experiencing food aversion due to taste and smell changes may be unable to respond to these agents. Of the appetite stimulants available for use in clinical practice only Marinol, or THC, has the potential to increase food intake by improving appetite as well as by amplifying the taste of food through the brain's reward pathway.

A 22-day, double blind, randomized, placebo-controlled trial will be conducted. Participants will start at 2.5mg of THC or placebo once daily for the first 3 days and then increase to 2.5mg of THC or placebo twice daily before lunch and supper. Participant's will complete the following survey tools pre and post-treatment: Taste and Smell Survey to assess the severity and change in chemosensory complaint scores; 3-day dietary record to determine the change in caloric intake and shift in food preference by macronutrient analysis; 24-hour urine collections to validate the 3-day dietary record; Satiety Labelled Intensity Magnitude scale for subjective appetite ratings; Food Preference Checklist to assess objective shifts in macronutrient and flavor preferences; Functional Assessment of Anorexia/Cachexia Therapy questionnaire to assess participant's QOL; interview to determine the cause and effects of chemosensory alterations; Edmonton Symptom Assessment Scale to assess nausea; and Side Effect Survey to document the tolerability of the drug (post-treatment only). Participants will complete the survey tools with the aid of the researcher. All tools are short and easy to complete, which minimizes patient burden.

ELIGIBILITY:
Inclusion Criteria:

* advanced cancer patients (defined as locally recurrent or metastatic) over 18 years old with a decreased food intake for at least 2 weeks (reported by physician or subject)
* able to complete questionnaires in English
* able to provide informed consent
* life expectancy of greater than 2 months (as determined by physician)
* chemosensory complaint score > 1

Exclusion Criteria:

* receiving enteral or parenteral feedings
* allergies or sensitivity to THC and/or sesame seed oil
* history of substance abuse or psychotic episodes
* mechanical obstruction of alimentary tract, mouth or nose
* received chemotherapy in the last 2 weeks
* received radiation therapy to the head/neck area
* brain tumor
* nausea score greater than 5 on ESAS
* history of tachyarrhythmias, angina pectoris or hypertension
* current diagnosis of liver impairment
* use of marijuana within 30 days prior to start of trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-08; Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Total caloric intake | 22 days

SECONDARY OUTCOMES:
self-perceived chemosensory ability | 22 days
palatable food intake | 22 days
self-perceived appetite | 22 days
changes in nausea | 22 days
safety and tolerability | 22 days

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid H. de Kock, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (2):
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Royal Victoria Hospital, Montreal, Quebec

REFERENCES:
- [Background] DeWys WD, Walters K. Abnormalities of taste sensation in cancer patients. Cancer. 1975 Nov;36(5):1888-96. doi: 10.1002/1097-0142(197511)36:53.0.co;2-y. PMID 1192373
- [Background] Jatoi A, Windschitl HE, Loprinzi CL, Sloan JA, Dakhil SR, Mailliard JA, Pundaleeka S, Kardinal CG, Fitch TR, Krook JE, Novotny PJ, Christensen B. Dronabinol versus megestrol acetate versus combination therapy for cancer-associated anorexia: a North Central Cancer Treatment Group study. J Clin Oncol. 2002 Jan 15;20(2):567-73. doi: 10.1200/JCO.2002.20.2.567. PMID 11786587
- [Background] Nelson K, Walsh D, Deeter P, Sheehan F. A phase II study of delta-9-tetrahydrocannabinol for appetite stimulation in cancer-associated anorexia. J Palliat Care. 1994 Spring;10(1):14-8. PMID 8035251
- [Derived] Brisbois TD, de Kock IH, Watanabe SM, Mirhosseini M, Lamoureux DC, Chasen M, MacDonald N, Baracos VE, Wismer WV. Delta-9-tetrahydrocannabinol may palliate altered chemosensory perception in cancer patients: results of a randomized, double-blind, placebo-controlled pilot trial. Ann Oncol. 2011 Sep;22(9):2086-2093. doi: 10.1093/annonc/mdq727. Epub 2011 Feb 22. PMID 21343383